CLINICAL TRIAL: NCT02906566
Title: Discovery of Effects of Retinol on Human Skin Aging in Individuals of East Asian Descent
Brief Title: Retinol on Human Skin Aging in East Asian Descent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne Chang, Associate Professor of Dermatology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 33762
Record Dates: First submitted 2016-02-26; First posted 2016-09-20 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Intrinsic Aging of Skin
MeSH Terms: interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Older Group Ages 55-75 (Other): Active and Placebo. Participants received retinol lotion on one arm and placebo to match on the other arm.
  Interventions: Drug: Retinol; Drug: Placebo
- Young Group Ages 18-25 (No Intervention): Participants in the group will give tissue sample only for comparison.

INTERVENTIONS:
Drug: Retinol — Retinol in the form of vitamin A lotion
  Arms: Older Group Ages 55-75
Drug: Placebo — Placebo of Retinol
  Arms: Older Group Ages 55-75

SUMMARY:
There has been increasing evidence for different rates of natural aging in humans and one of the best organs to study human aging is skin. Studies have demonstrated anti-aging effects of topical agents (such as creams, gels, lotions, or ointments) and one of them, retinol or vitamin A, was shown to decrease fine wrinkling in skin of older individuals. Additionally, studies of retinol in humans have largely occurred in white populations and so this study aims to focus on skin aging in individuals of East Asian descent as they represent a majority of the world population. This study aims to better characterize the molecular basis of rejuvenation effects and to potentially discover new topical agents with similar and/or more effective preservation of skin youthfulness.

ELIGIBILITY:
Inclusion Criteria:

* able to provide written informed consent
* older group: age between 50 and 75 years
* young group: age 18 to 25 years
* all four grandparents of Han Chinese, Japanese, Korean descent
* body mass index within normal or overweight range
* no history of weight loss of >20 lbs within past 5 years

Exclusion Criteria:

* skin condition in the areas of skin biopsy that would obscure results of analysis
* topical creams or treatment to arms 2 weeks prior to study baseline visit
* individuals with known hypersensitivity to retinoid class of agents (older group only)
* prior anti-aging treatments to arms including retinol, microdermabrasion within 2 weeks of baseline visit
* prior laser therapy or surgical procedure to arms
* prior radiation or other trauma (extensive burns or abrasions) to arm skin
* hormone-based therapy within 4 weeks of enrollment

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Dermatology, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 110 participants were consented; 34 participants were assigned to a study arm.
Units Other Than Participants: Arms
Groups:
- Older Group Ages 55-75: Participants received retinol lotion on one arm and placebo to match on the other arm.
- Young Group Ages 18-25: Participants in the group will give a tissue sample from one arm only for comparison.
Period: Overall Study
Arm/Group | Older Group Ages 55-75 | Young Group Ages 18-25
Started | 24; 48 Arms | 10; 10 Arms
Completed | 21; 42 Arms | 10; 10 Arms
Not Completed | 3; 6 Arms | 0; 0 Arms

BASELINE CHARACTERISTICS:
Population: Participants who were assigned to a treatment arm were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Group Ages 55-75 | Young Group Ages 18-25 | Total
Number analyzed (Participants) | 24 | 10 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 13 | 0 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (4.7) | 21.7 (3.1) | 51.7 (21.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 10 | 34
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 10 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Genes Upregulated or Downregulated as Assessed by RNA Sequencing (Older Group, Retinol Versus Placebo)
Description: Differences in transcript levels are reported as the number that were upregulated or downregulated in the participant's retinol-treated arm versus their placebo-treated arm.
Time Frame: Week 12
Population: Participants in the "Young Group Ages 18-25" attended a single study visit at week 1 to provide tissue samples for comparison purposes, and are not included in this analysis.
Measure: Number; unit: genes
Units Other Than Participants: genes
Arm/Group | Older Group Ages 55-75
Number analyzed (Participants) | 24
Number analyzed (genes) | 56615
genes
  Upregulated | 23
  Downregulated | 21

2. Secondary Outcome: Transepidermal Water Loss
Description: Transepidermal Water Loss of arm skin was measured in units of grams/hours/meters squared.
Time Frame: Baseline; Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/h/m^2
Groups:
- Retinol Treated Arm: Participants in the older group (ages 55-75), retinol arm.
- Placebo Treated Arm: Participants in the older group (ages 55-75), placebo arm.
Arm/Group | Retinol Treated Arm | Placebo Treated Arm
Number analyzed (Participants) | 21 | 21
g/h/m^2
  Baseline | 17.1 (10.2) | 16.2 (11.7)
  Week 12 | 9.4 (6.7) | 10.2 (6.1)

3. Secondary Outcome: Severity of Arm Skin Wrinkling
Description: Wrinkling was assessed by the investigator using a 10-point Likert scale (range 0 to 9, lower scores correspond to less wrinkling).
Time Frame: Baseline; Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Retinol Treated Arm | Placebo Treated Arm
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline | 5.15 (1.96) | 5.5 (1.59)
  Week 12 | 4.85 (1.79) | 5.175 (1.28)

4. Secondary Outcome: Elasticity on Arm Skin
Description: Elasticity was assessed using cutometry (R2 curve) as millimeters per second
Time Frame: Baseline; week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters per second
Arm/Group | Retinol Treated Arm | Placebo Treated Arm
Number analyzed (Participants) | 21 | 21
millimeters per second
  Baseline | 0.8623 (0.0791) | 0.8753 (0.0464)
  Week 12 | 0.8587 (0.0655) | 0.8576 (0.0684)

5. Secondary Outcome: Count of Participants With Skin and Subcutaneous Adverse Events as a Measure of Type and Severity of Adverse Events
Description: Skin and subcutaneous adverse events were assessed for this outcome and documented and scored according to CTCAE version 4.03.
Time Frame: Baseline through week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Retinol Treated Arm | Placebo Treated Arm
Number analyzed (Participants) | 21 | 21
Participants
  Dermatitis (Grade 1) | 1 | 1
  Tingling sensation after application (Grade 1) | 0 | 1

6. Primary Outcome: Number of Genes Upregulated or Downregulated as Assessed by RNA Sequencing (Younger Group Versus Older Group as Baseline)
Description: Differences in transcript levels are reported as the number of genes that were upregulated or downregulated in the Younger Group participant tissue samples, as compared to a baseline provided by tissue samples collected from the Older Group (prior to their treatment).
Time Frame: Week 1
Population: Only the participants in "Younger Group (ages 18-25)" are included in the analysis, since a comparison of the baseline data for the "Older Group (ages 55-75)" against itself is not clinically meaningful.
Measure: Number; unit: genes
Units Other Than Participants: genes
Arm/Group | Young Group Ages 18-25
Number analyzed (Participants) | 10
Number analyzed (genes) | 56615
genes
  Downregulated | 775
  Upregulated | 587

ADVERSE EVENTS:
Time Frame: Up to 12 weeks.
Arm/Group | Older Group Ages 55-75 | Young Group Ages 18-25
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/10
Other Adverse Events (participants affected / at risk) | 4/24 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Group Ages 55-75 (N=24) | Young Group Ages 18-25 (N=10)
Upper respiratory infection (Infections and infestations) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT02906566/Prot_SAP_000.pdf